CLINICAL TRIAL: NCT06284655
Title: The Effect of a Brief Educational Intervention for Adults With ADHD: a Randomized Control Trial
Brief Title: The Effect of a Brief Educational Intervention for Adults With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 635362 a
Record Dates: First submitted 2023-12-01; First posted 2024-02-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: ADHD
Keywords: ADHD; patient education; psychoeducation; patients' satisfaction; general self-efficacy; self-management; self-management skills; group-based education; peer co-led
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel two-arms randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Blinded statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Experimental): Patients randomized to the intervention group will start with peer co-led group-based psychoeducation, combined with digital video- and written information.
  Interventions: Behavioral: group-based combined with innovative technology education
- Control group (Active Comparator): The control group will receive treatment as usual after randomization
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: group-based combined with innovative technology education — The intervention combines brief group-based psychoeducation, and digital video- and written information, to deliver an early self-management educational program. The intervention introduces a group-breaking approach, featuring a self-managed peer co-led educational group, in collaboration with user representatives from Vårres and the ADHD organisation. This patient-centred educational programme covers crucial topics such as self-help tools, treatment options and experiences, patients' rights, and self-management, in addition to treatment as usual.
  Other Names: Treatment as usual
  Arms: Educational intervention
Other: Standard treatment — Treatment as usual.
  Arms: Control group

SUMMARY:
This RCT-study proposes the evaluation of an intensive educational intervention tailored for adults with Attention Deficit Hyperactivity Disorder (ADHD) in community mental health centers (CMHCs). Given the prevalent challenges of prolonged waiting lists and low patient engagement in CMHCs, the research seeks to assess the efficacy of this intervention in enhancing patient engagement, self-efficacy, satisfaction with the information and overall health outcomes. The intervention, developed collaboratively with user representatives, combines a brief group-based educational sessions with standard clinical care. The primary hypotheses posit that this approach will lead to increased patient satisfaction with the treatment, patient self-efficacy, and activation compared to conventional treatment. Additionally, it aims to improve patients' satisfaction with information received. The study will employ a ITT analysis to assess the intervention's effects against usual treatment practices in outpatient settings. The anticipated outcome is a significant improvement in level of patient satisfaction, level of self-efficacy and level of satisfaction with the received information for patients with ADHD, potentially informing clinical practices and optimizing care for adults with ADHD.

DETAILED DESCRIPTION:
Community mental health centres (CMHCs) face significant challenges in meeting the needs of individuals with mental health issues. For example, due to high demand there are long waiting lists and low engagement rates. To address these challenges, innovative interventions are urgently needed to improve patient engagement, coping skills, and overall health outcomes. Educational and self-management interventions have shown promise in enhancing patient satisfaction and patient activation in other contexts and may therefore be potential solutions to reduce the identified challenges in the mental health service. To bridge these knowledge and practice gaps, this application proposes the evaluation of one educational intervention tailored specifically for adults with ADHD. This intervention aims to enhance patient engagement, treatment satisfaction, activation and overall outcomes.

The main hypotheses are that the new educational approach, developed in cooperation with user representatives, will result in higher patient engagement, increase patient satisfaction with the treatment, self-efficacy and patient activation.

The researchers hypothesized that the new educational intervention, through a brief group-based approach and in conjunction with standard clinical care, will improve patients' satisfaction, patients' self-efficacy, satisfaction with the information, as well as patient activation, compared to the usual treatment, in outpatient mental health settings.

This intervention has the potential to empower patients, increase their engagement in treatment, and improve their overall functioning. By demonstrating the efficacy of this approach, this research will inform clinical practice and contribute to the optimization of care for adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed ADHD-diagnosis
* Speaking a Scandinavian language
* Willing to participate

Exclusion Criteria:

* Unable to give informed consent
* In-patient on a acute psychiatric ward
* Severe learning difficulties
* Involvement in other research studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in client satisfaction using CSQ | After the intervention up to 4 weeks [post intervention] and up to 56 weeks [follow up]
  Client satisfaction will be measured with Client Satisfaction Questionnaire 4 items (CSQ4). Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction), with higher scores indicating greater satisfaction.
Change in general self-efficacy using GSE-6 | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  General Self-Efficacy Scale is a 6-item scale with answers ranging from 1 ('not at all true') to 4 ('exactly true'). Total scores range from 6 to 24, with higher scores indicating greater self-efficacy.
Change in satisfaction with the information | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  The satisfaction with the information survey includes 3 items, which score from 1 (not satisfied) to 5 (very satisfied), the option (I don't know) gives 0 points. The total score ranges from 3 to 15, with higher scores indicating higher satisfaction with the information
Knowledge and treatment preferences | At baseline, 1 week before the intervention [pre-intervention], and at 4 weeks [post intervention]
  Knowledge will be measured by five questions answered on six-point ordinary scale, and one question answered as "yes", "no", "don't know"

SECONDARY OUTCOMES:
Change in patient activation using PAM | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Patient activation will be measured with the Norwegian version of the Patient Activation Measure (PAM), which consists of 13 items, and total score ranges from 0 to 100, higher total score indicates higher patient activation
Change in ADHD-related symptoms using ASRS | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  ADHD specific subscale and the ADHD Self-Report Scale (ASRS). Each item is answered on a five point scale ranging from 0 ("never") to 4 ("very often"). Higher scores indicates more pronounced symptoms.
Change in ADHD-related symptoms using SCL-9 | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Hopkin's Symptoms Checklist 9-items (SCL-9), consists of nine items scored from 0 ("not at all") to 4 ("very much"), and the possible total score ranges from 0 to 36. The higher score in SCL-9 indicates more pronounced symptoms of the disorder.
Change in depression and anxiety symptoms using PHQ-4 | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Patient Health Questionnaire for Depression and Anxiety (PHQ-4), consists of 4 items. Two questions assess anxiety symptoms, and two questions assess depression symptoms. Possible answers are given by a four-point scale ranging from "not at all" (0) to "nearly every day" (3), making a possible score range of 0-12. A higher score represents higher symptom severity.
Change in patient enablement using PEN-13 | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Patient Enablement-13 have 13 items. items are graded on a five/point scale and values can range from 13 (minimum enablement) to 65 points (maximum enablement).
Change in stress level using PSS-4 | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Perceived Stress Scale 4 (PSS-4), consists of 4 items. All items are rated on an ordinal 5-point scale, coded 0 through 4, and total score ranges from 0 to 16 where a higher score represents a higher subjective stress level.
Change in level of functioning using WSAS | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Work and Social Adjustment scale (WSAS) consists of 5 items with the range from 0 (not at all) to 8 (very severely), with the total score from 0 to 40, where the higher score indicates more severe functional impairments.
Change in ADHD Quality of life using AAQoL | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Quality of life was measured using the Adult ADHD quality of life scale (AAQoL). The AAQoL consists of 29 questions. Each item is rated on a 1 to 5 Likert scale. The total score ranges from 0 to 100. A higher score indicates higher quality of life.
Change in Health-related Quality of life using EQ-5D-5L | At baseline, 1 week before the intervention [pre-intervention], at 4 weeks [post intervention] and up to 56 weeks [follow up]
  Quality of life was measured using the 5-level EQ-5D scale (EQ-5D-5L), which consists of 5 questions, that range on 5-point scale, which reflect the level of the dimension of the functions. Higher score indicates worse quality of life.

OTHER OUTCOMES:
Cost | Up to 56 weeks [follow up]
  Cost development to evaluate its cost-benefit
Health care usage | Up to 56 weeks [follow up]
  Data from official patient register will be used (drop out, number of consultations, type of treatment, length of treatment, attendance rates and diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Loreto Lara-Cabrera, PhD, Principal Investigator — Norwegian University of Science and Technology; Rolf W. Gråwe, PhD, Prof., Study Chair — Norwegian University of Science and Technology; Liv S. Engvik, Cand Psychol, Study Chair — St. Olavs Hospital
Locations (1):
- St Olav's Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No